CLINICAL TRIAL: NCT00626600
Title: An Open, Multi-centre, Non-comparative Observational Study to Assess the Safety and Tolerability of Oxycodone Injection 50 mg/mL as a Subcutaneous Infusion in Patients With Severe Cancer Pain.
Brief Title: A Study to Assess the Safety and Tolerability of Oxycodone Hydrochloride 50mg/mL Administered as an Infusion
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXI3001; 2007-005101-21
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Severe Caner Pain
Keywords: Oxycodone Hydrochloride 50mg/mL; Observational; Infusion; Severe cancer pain
MeSH Terms: conditions — Cancer Pain | interventions — Oxycodone

INTERVENTIONS:
Drug: Oxycodone Hydrochloride

SUMMARY:
Assessing the safety and tolerability of Oxycodone Hydrochloride 50mg/mL in subjects with severe cancer pain.

DETAILED DESCRIPTION:
This is study involving a treatment phase of up to 20 days. During this time patients will receive Oxycodone Hydrochloride 50mg/ml as a subcutaneous infusion. During the treatment phase, safety will be assessed by documentation of type and frequency of spontaneously reported adverse events and adverse events noted after assessment of the infusion site (every 24 hours and when resited). The subjects will be followed up for 7 days to collect information on ongoing AEs/SAEs and any new AEs/SAEs that may have occurred.

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects aged 18 years and above, who have severe cancer pain.
2. Subjects who require a strong opioid by subcutaneous infusion to stabilise and manage their cancer pain effectively.
3. Subjects who give written informed consent to participate in the study.
4. Subjects who agree to their primary care physician being informed of their participation in the study.
5. Subjects who consent to processing of their trial data according to the requirements of the UK Data Protection Act 1998.

Exclusion Criteria

1. Subjects who are pregnant, lactating or in the Investigators opinion are at risk of conceiving and are not using adequate contraception measures.
2. Subjects with known hypersensitivity (allergic reaction) to oxycodone, any other opioids or any of the excipients.
3. Subjects who are planned to receive chemotherapy during the study treatment period or are currently receiving continuous i.v. chemotherapy infusion.
4. Subjects with neutropenia, thrombocytopenia or coagulation disorders.
5. Subjects with any contraindications to oxycodone as outlined in the Investigator Brochure or Summary Product Information sheet for oxycodone.
6. Subjects who are currently participating in another clinical research study involving a new chemical entity.
7. Subjects whom the Investigator believes to be medically unfit to receive the study medication, or unsuitable for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of Oxycodone hydrochloride injection 50 mg/mL | 20 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden Hospital, London, United Kingdom

REFERENCES:
- See also: Link to Results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=OXI3001